CLINICAL TRIAL: NCT03992625
Title: Clinical Outcomes for Deep Brain Stimulation for Parkinson Disease, Tremor, and Dystonia
Brief Title: Clinical Outcomes for Deep Brain Stimulation
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Mwiza Ushe, Assistant Professor, Washington University School of Medicine
Other Study IDs: 201101744; R01NS075321 (NIH); R01NS097437 (NIH); R21NS098020 (NIH); T32EB021955 (NIH)
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia
Keywords: Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Deep Brain Stimulation — High frequency electrical stimulation of deep brain nuclei for the treatment of movement disorders

SUMMARY:
The object of this study is to longitudinally collect clinical outcomes of patients receiving deep brain stimulation for movement disorders with the objective of making retrospective comparisons and tracking of risks, benefits, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Levodopa responsive Parkinson disease OR
* Medically refractory Essential Tremor OR
* Medically refractory Dystonia

Exclusion Criteria:

* Dementia (Mattis Dementia Rating Scale <130)
* Structural abnormalities precluding intracranial surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving deep brain stimulation for movement disorders
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-01-03 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
UPDRS | Change in UPDRS at 1 year after DBS (from preoperative baseline).
  United Parkinson's Disease Rating Scale (global assessment of motor, non-motor, and quality of life associated with symptoms of Parkinson disease). Total scores range from 0-199. Particular emphasis is paid to subsection 3 (motor), where scores range from 0-56.

CONTACTS AND LOCATIONS:
Overall Officials: Mwiza Ushe, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No